CLINICAL TRIAL: NCT07163767
Title: Acute Myocardial Infarction Prediction Using Artificial Intelligence Applied to Electrocardiogram Images
Status: Active, not recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Liu yong, Professor, Guangdong Provincial People's Hospital
Other Study IDs: KY2025-514
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Acute Myocardial Infarction (AMI); Electrocardiography; Artifical Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiorenal ImprovemeNt II (CIN-II): This is a multi-center, retrospective observation study collecting data on 184855 coronary angiography patients from January 2000 to Decemeber 2020.
  Interventions: Other: Deep learning approach of ECG for AMI detection

INTERVENTIONS:
Other: Deep learning approach of ECG for AMI detection — AMIdECG was trained to perform AMI detection in a supervised manner as a classification task. And the classification labels of AMI subtypes (" STEMI "or" NSTEMI ") or non-AMI states used during the training phase are real-world diagnostic results

SUMMARY:
The goal of this observational study is to develop and validate an artificial intelligence(AI)-based prediction model for new-onset acute myocardial infarction(AMI) using electrocardiogram(ECG) data. The main question it aims to answer is whether the AI-based ECG accurately forecast new-onset AMI by previous ECG data with 'normal' diagnosis?

DETAILED DESCRIPTION:
Myocardial infarction (MI), as one of the most critical acute clinical events in cardiovascular diseases, has high morbidity and mortality, imposing a significant burden on public health and medical resources. Traditional risk assessment for MI relies on clinical indicators (e.g., lipids, blood pressure, diabetes status, family history) and cardiac imaging, but these methods often suffer from invasive procedure, high cost, or limited predictive accuracy. Electrocardiography (ECG), a non-invasive, widely available, and low-cost modality, captures rich electrophysiological signals reflecting cardiac function. However, conventional analysis methods struggle to detect subtle, progressive patterns in ECG signals, leading to sub-optimal sensitivity and specificity in predicting new-onset MI.

Recent advancements in deep learning and big data have enabled significant progress in ECG-based prediction models. For example, deep convolutional neural networks (CNNs) for automatic feature extraction and pattern recognition from 12-lead ECGs have demonstrated promise in predicting cardiovascular events such as atrial fibrillation, left ventricular hypertrophy, and heart failure re-hospitalization. AI algorithms have also been shown to extract subtle information from ECGs that traditional methods miss, such as dynamic changes in ventricular electrical activity and early signs of micro-myocardial injury, enabling early risk warning of cardiac events. While numerous ECG-based AI models exist for predicting arrhythmia , heart failure, and other cardiovascular outcomes, research on predicting new-onset MI-particularly using non-invasive ECG data and deep learning to extract latent predictive markers-remains in its infancy. Traditional risk models, though successful in MI prevention, lack precision in individual-level prediction and early intervention.

This study aims to leverage large-scale electronic health records and ECG datasets with advanced deep learning to explore the quantitative relationship between fine-grained ECG signal features and MI incidence, thereby developing a clinical tool for early risk assessment. Inspirations also derive from recent attempts to build multi-modal prediction models combining ECG with physiological, genetic, and biochemical markers. Additionally, studies have highlighted ECG's unique advantages in evaluating myocardial compensatory mechanisms and early injury. Despite existing ECG-AI applications, direct prediction of new-onset MI remains a critical unmet need and a key direction for precision medicine using AI.

This is a multi-center observational cohort study. Large-scale in-hospital ECG data will be integrated to develop a deep learning model for MI prediction using an end-to-end deep neural network approach, with the goal of deriving a high-performance model for new-onset MI prediction. The ECG data from 5 multicenter Cardiorenal ImprovemeNt II (CIN-II) sites between 2010-2023 will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in cardiology department with myocardial injury marker testing (troponin T/I).
* In-hospital patients with ECG records.

Exclusion Criteria:

* First ECG obtained in emergency department.
* ACS diagnosis within 1 month of first ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In-hospital patients with ECG records
Sampling Method: Non-Probability Sample
Enrollment: 150000 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute myocardial infarction (AMI) | From June 2025 to April 2026
  AMI was defined as STEMI, NSTEMI using ICD-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadasivuni S, Saha M, Bhatia N, Banerjee I, Sanyal A. Fusion of fully integrated analog machine learning classifier with electronic medical records for real-time prediction of sepsis onset. Sci Rep. 2022 Apr 5;12(1):5711. doi: 10.1038/s41598-022-09712-w. PMID 35383233
- [Background] Jawade P, Khillare KM, Mangudkar S, Palange A, Dhadwad J, Deshmukh M. A Comparative Study of Ischemia-Modified Albumin: A Promising Biomarker for Early Detection of Acute Coronary Syndrome (ACS). Cureus. 2023 Aug 30;15(8):e44357. doi: 10.7759/cureus.44357. eCollection 2023 Aug. PMID 37779796
- [Background] Swenne CA, Ter Haar CC. Context-independent identification of myocardial ischemia in the prehospital ECG of chest pain patients. J Electrocardiol. 2024 Jan-Feb;82:34-41. doi: 10.1016/j.jelectrocard.2023.10.009. Epub 2023 Nov 7. PMID 38006762
- [Background] Akbilgic O, Butler L, Karabayir I, Chang PP, Kitzman DW, Alonso A, Chen LY, Soliman EZ. ECG-AI: electrocardiographic artificial intelligence model for prediction of heart failure. Eur Heart J Digit Health. 2021 Oct 9;2(4):626-634. doi: 10.1093/ehjdh/ztab080. eCollection 2021 Dec. PMID 34993487
- [Background] Aufiero S, Bleijendaal H, Robyns T, Vandenberk B, Krijger C, Bezzina C, Zwinderman AH, Wilde AAM, Pinto YM. A deep learning approach identifies new ECG features in congenital long QT syndrome. BMC Med. 2022 May 3;20(1):162. doi: 10.1186/s12916-022-02350-z. PMID 35501785
- [Background] Serhal H, Abdallah N, Marion JM, Chauvet P, Oueidat M, Humeau-Heurtier A. Overview on prediction, detection, and classification of atrial fibrillation using wavelets and AI on ECG. Comput Biol Med. 2022 Mar;142:105168. doi: 10.1016/j.compbiomed.2021.105168. Epub 2022 Jan 1. PMID 35033876
- [Background] Elul Y, Rosenberg AA, Schuster A, Bronstein AM, Yaniv Y. Meeting the unmet needs of clinicians from AI systems showcased for cardiology with deep-learning-based ECG analysis. Proc Natl Acad Sci U S A. 2021 Jun 15;118(24):e2020620118. doi: 10.1073/pnas.2020620118. PMID 34099565
- [Background] Liu YL, Lin CS, Cheng CC, Lin C. A Deep Learning Algorithm for Detecting Acute Pericarditis by Electrocardiogram. J Pers Med. 2022 Jul 15;12(7):1150. doi: 10.3390/jpm12071150. PMID 35887647
- [Background] Pignolo RJ. AI-ECG and the Prediction of Accelerated Aging. Mayo Clin Proc. 2023 Apr;98(4):502-503. doi: 10.1016/j.mayocp.2023.02.016. No abstract available. PMID 37019510
- [Background] Wang X, Khurshid S, Choi SH, Friedman S, Weng LC, Reeder C, Pirruccello JP, Singh P, Lau ES, Venn R, Diamant N, Di Achille P, Philippakis A, Anderson CD, Ho JE, Ellinor PT, Batra P, Lubitz SA. Genetic Susceptibility to Atrial Fibrillation Identified via Deep Learning of 12-Lead Electrocardiograms. Circ Genom Precis Med. 2023 Aug;16(4):340-349. doi: 10.1161/CIRCGEN.122.003808. Epub 2023 Jun 6. PMID 37278238
- [Background] Attia ZI, Friedman PA. Explainable AI for ECG-based prediction of cardiac resynchronization therapy outcomes: learning from machine learning? Eur Heart J. 2023 Feb 21;44(8):693-695. doi: 10.1093/eurheartj/ehac733. No abstract available. PMID 36546617
- [Background] Martinez-Selles M, Marina-Breysse M. Current and Future Use of Artificial Intelligence in Electrocardiography. J Cardiovasc Dev Dis. 2023 Apr 17;10(4):175. doi: 10.3390/jcdd10040175. PMID 37103054
- [Background] Butler L, Ivanov A, Celik T, Karabayir I, Chinthala L, Tootooni MS, Jaeger BC, Patterson LT, Doerr AJ, McManus DD, Davis RL, Herrington D, Akbilgic O. Time-Dependent ECG-AI Prediction of Fatal Coronary Heart Disease: A Retrospective Study. J Cardiovasc Dev Dis. 2024 Dec 8;11(12):395. doi: 10.3390/jcdd11120395. PMID 39728285
- [Background] Sekhri N, Feder GS, Junghans C, Hemingway H, Timmis AD. How effective are rapid access chest pain clinics? Prognosis of incident angina and non-cardiac chest pain in 8762 consecutive patients. Heart. 2007 Apr;93(4):458-63. doi: 10.1136/hrt.2006.090894. Epub 2006 Jun 21. PMID 16790531
- [Background] Stubbs P, Collinson P, Moseley D, Greenwood T, Noble M. Prospective study of the role of cardiac troponin T in patients admitted with unstable angina. BMJ. 1996 Aug 3;313(7052):262-4. doi: 10.1136/bmj.313.7052.262. PMID 8704534
- [Background] Farkouh ME, Smars PA, Reeder GS, Zinsmeister AR, Evans RW, Meloy TD, Kopecky SL, Allen M, Allison TG, Gibbons RJ, Gabriel SE. A clinical trial of a chest-pain observation unit for patients with unstable angina. Chest Pain Evaluation in the Emergency Room (CHEER) Investigators. N Engl J Med. 1998 Dec 24;339(26):1882-8. doi: 10.1056/NEJM199812243392603. PMID 9862943
- [Background] Fox KA, Goodman SG, Klein W, Brieger D, Steg PG, Dabbous O, Avezum A. Management of acute coronary syndromes. Variations in practice and outcome; findings from the Global Registry of Acute Coronary Events (GRACE). Eur Heart J. 2002 Aug;23(15):1177-89. doi: 10.1053/euhj.2001.3081. PMID 12127920
- [Background] Grech ED, Ramsdale DR. Acute coronary syndrome: unstable angina and non-ST segment elevation myocardial infarction. BMJ. 2003 Jun 7;326(7401):1259-61. doi: 10.1136/bmj.326.7401.1259. No abstract available. PMID 12791748
- [Background] Pollack CV Jr, Sites FD, Shofer FS, Sease KL, Hollander JE. Application of the TIMI risk score for unstable angina and non-ST elevation acute coronary syndrome to an unselected emergency department chest pain population. Acad Emerg Med. 2006 Jan;13(1):13-8. doi: 10.1197/j.aem.2005.06.031. Epub 2005 Dec 19. PMID 16365321
- [Background] Sinha MK, Roy D, Gaze DC, Collinson PO, Kaski JC. Role of "Ischemia modified albumin", a new biochemical marker of myocardial ischaemia, in the early diagnosis of acute coronary syndromes. Emerg Med J. 2004 Jan;21(1):29-34. doi: 10.1136/emj.2003.006007. PMID 14734370
- [Background] de Beer FC, Hind CR, Fox KM, Allan RM, Maseri A, Pepys MB. Measurement of serum C-reactive protein concentration in myocardial ischaemia and infarction. Br Heart J. 1982 Mar;47(3):239-43. doi: 10.1136/hrt.47.3.239. PMID 7059401
- [Background] Katus HA, Remppis A, Neumann FJ, Scheffold T, Diederich KW, Vinar G, Noe A, Matern G, Kuebler W. Diagnostic efficiency of troponin T measurements in acute myocardial infarction. Circulation. 1991 Mar;83(3):902-12. doi: 10.1161/01.cir.83.3.902. PMID 1999039
- [Background] Yagi R, Goto S, Himeno Y, Katsumata Y, Hashimoto M, MacRae CA, Deo RC. Artificial intelligence-enabled prediction of chemotherapy-induced cardiotoxicity from baseline electrocardiograms. Nat Commun. 2024 Mar 21;15(1):2536. doi: 10.1038/s41467-024-45733-x. PMID 38514629
- [Background] Shen CP, Muse ED. Towards an artificial intelligence-augmented, ECG-enabled physical exam. Lancet Digit Health. 2022 Feb;4(2):e78-e79. doi: 10.1016/S2589-7500(21)00281-8. Epub 2022 Jan 5. No abstract available. PMID 34998739
- [Background] Lincoff AM, Brown-Frandsen K, Colhoun HM, Deanfield J, Emerson SS, Esbjerg S, Hardt-Lindberg S, Hovingh GK, Kahn SE, Kushner RF, Lingvay I, Oral TK, Michelsen MM, Plutzky J, Tornoe CW, Ryan DH; SELECT Trial Investigators. Semaglutide and Cardiovascular Outcomes in Obesity without Diabetes. N Engl J Med. 2023 Dec 14;389(24):2221-2232. doi: 10.1056/NEJMoa2307563. Epub 2023 Nov 11. PMID 37952131
- [Background] Dhingra LS, Aminorroaya A, Sangha V, Pedroso AF, Asselbergs FW, Brant LCC, Barreto SM, Ribeiro ALP, Krumholz HM, Oikonomou EK, Khera R. Heart failure risk stratification using artificial intelligence applied to electrocardiogram images: a multinational study. Eur Heart J. 2025 Mar 13;46(11):1044-1053. doi: 10.1093/eurheartj/ehae914. PMID 39804243
- [Background] Biscaglia S, Guiducci V, Escaned J, Moreno R, Lanzilotti V, Santarelli A, Cerrato E, Sacchetta G, Jurado-Roman A, Menozzi A, Amat Santos I, Diez Gil JL, Ruozzi M, Barbierato M, Fileti L, Picchi A, Lodolini V, Biondi-Zoccai G, Maietti E, Pavasini R, Cimaglia P, Tumscitz C, Erriquez A, Penzo C, Colaiori I, Pignatelli G, Casella G, Iannopollo G, Menozzi M, Varbella F, Caretta G, Dudek D, Barbato E, Tebaldi M, Campo G; FIRE Trial Investigators. Complete or Culprit-Only PCI in Older Patients with Myocardial Infarction. N Engl J Med. 2023 Sep 7;389(10):889-898. doi: 10.1056/NEJMoa2300468. Epub 2023 Aug 26. PMID 37634150
- [Background] Kromhout D, Giltay EJ, Geleijnse JM; Alpha Omega Trial Group. n-3 fatty acids and cardiovascular events after myocardial infarction. N Engl J Med. 2010 Nov 18;363(21):2015-26. doi: 10.1056/NEJMoa1003603. Epub 2010 Aug 28. PMID 20929341
- [Background] Dupulthys S, Dujardin K, Anne W, Pollet P, Vanhaverbeke M, McAuliffe D, Lammertyn PJ, Berteloot L, Mertens N, De Jaeger P. Single-lead electrocardiogram Artificial Intelligence model with risk factors detects atrial fibrillation during sinus rhythm. Europace. 2024 Feb 1;26(2):euad354. doi: 10.1093/europace/euad354. PMID 38079535
- [Background] Nechita LC, Nechita A, Voipan AE, Voipan D, Debita M, Fulga A, Fulga I, Musat CL. AI-Enhanced ECG Applications in Cardiology: Comprehensive Insights from the Current Literature with a Focus on COVID-19 and Multiple Cardiovascular Conditions. Diagnostics (Basel). 2024 Aug 23;14(17):1839. doi: 10.3390/diagnostics14171839. PMID 39272624
- [Background] Chen HY, Lin CS, Fang WH, Lee CC, Ho CL, Wang CH, Lin C. Artificial Intelligence-Enabled Electrocardiogram Predicted Left Ventricle Diameter as an Independent Risk Factor of Long-Term Cardiovascular Outcome in Patients With Normal Ejection Fraction. Front Med (Lausanne). 2022 Apr 11;9:870523. doi: 10.3389/fmed.2022.870523. eCollection 2022. PMID 35479951
- [Background] Lee HS, Kang S, Jo YY, Son JM, Lee MS, Kwon JM, Kim KH. AI-Enabled Smartwatch ECG: A Feasibility Study for Early Prediction and Prevention of Heart Failure Rehospitalization. JACC Basic Transl Sci. 2025 Mar;10(3):250-252. doi: 10.1016/j.jacbts.2025.01.005. Epub 2025 Feb 11. No abstract available. PMID 40139860
- [Background] Khurshid S, Friedman S, Reeder C, Di Achille P, Diamant N, Singh P, Harrington LX, Wang X, Al-Alusi MA, Sarma G, Foulkes AS, Ellinor PT, Anderson CD, Ho JE, Philippakis AA, Batra P, Lubitz SA. ECG-Based Deep Learning and Clinical Risk Factors to Predict Atrial Fibrillation. Circulation. 2022 Jan 11;145(2):122-133. doi: 10.1161/CIRCULATIONAHA.121.057480. Epub 2021 Nov 8. PMID 34743566